CLINICAL TRIAL: NCT02825056
Title: Comparison of Postoperative Hemodynamics After High Spinal Block With or Without Intrathecal Morphine in Cardiac Surgeries.
Brief Title: Postoperative Hemodynamics Comparison After High Spinal Block With or Without Intrathecal Morphine.
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, IMRAN HUSSAIN BHAT, Post operative hemodynamic investigator, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: NK/2676/DM/397
Record Dates: First submitted 2016-06-19; First posted 2016-07-07 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Vasoplegia
MeSH Terms: conditions — Vasoplegia | interventions — Bupivacaine; Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bupivacaine (Active Comparator): Intrathecal 8 ml single dose of 0.5% heavy Bupivacaine (Anawin heavy 0.5%).
  Interventions: Drug: Bupivacaine
- Bupivacaine + Morphine (Experimental): Intrathecal 8 ml single dose of 0.5% heavy Bupivacaine (Anawin heavy 0.5%) and 250 microgram of preservative free Morphine (VERMOR).
  Interventions: Drug: Bupivacaine + Morphine

INTERVENTIONS:
Drug: Bupivacaine — Intrathecal local anesthetic drug,Bupivacaine will be delivered in L3-L4 space.
  Other Names: Anawin heavy 0.5%,Neon laboratories LTD, Thane, India.
  Arms: Bupivacaine
Drug: Bupivacaine + Morphine — Intrathecal local anesthetic drug,Bupivacaine and Morphine will be delivered in L3-L4 space.
  Other Names: Anawin heavy 0.5%,and VERMOR 15,Verve, Delhi, India
  Arms: Bupivacaine + Morphine

SUMMARY:
There is paucity of literature on the effects of intrathecal morphine on the postoperative hemodynamics in the cardiac-surgical patients.We planned this study to compare the post-operative hemodynamic effects (particularly the incidence of vasoplegia in the two study groups) and outcome of combined general anesthesia + high spinal block, with or without intrathecal morphine in patients undergoing cardiac-surgical procedures in our set up.

DETAILED DESCRIPTION:
Introduction Currently various strategies are being developed for fast tracking in cardiac anaesthesia that includes use of shorter acting opioids , combined thoracic epidural or high spinal anaesthesia with GA, awake cardiac surgery along with normothermic or mild hypothermic cardiopulmonary bypass (CPB) and off pump surgeries. The aim of fast tracking is early extubation, early mobilization, decreased length of ICU and overall hospital stay, not only to reduce costs and human resource utilisation but also to reduce the postoperative morbidity and mortality while enhancing the quality of health care.

Traditionally high dose opioid anaesthesia has been used to abolish this stress response, however, some studies have shown that this technique of anaesthesia only relatively minimizes the stress response and does not completely block it.

Regional anaesthesia in the form of thoracic epidural anaesthesia (TEA) alone (awake cardiac anaesthesia) or combined with general anaesthesia (GA) has been used in cardiac surgical patients. One of the useful alternatives to TEA would be high spinal anaesthesia as the risk of haematoma associated with this procedure is much less than the epidural in cardiac surgical patients. The use of spinal anaesthesia in cardiac patients, particularly patients with stenotic valvular lesions has been for long viewed with much apprehension, primarily due to the perceived risk of hypotension as a result of sympatholysis. However, various studies using high spinal up to T1 level have proved such apprehensions to be invalid in the setting of cardiac surgery where patients are monitored intensively with invasive monitors and the hypotension managed at the earliest with the use of small aliquots or continuous infusion of vasoactive agents such as phenylephrine, norepinephrine, epinephrine, mephentermine as per the requirements of underlying cardiac lesion.

Although thoracic epidural anaesthesia has been studied and practiced, there is paucity of literature on the effects of intrathecal morphine on the postoperative hemodynamics in the cardiac-surgical patients.Hence, the investigators planned this study to compare the post-operative hemodynamic effects and outcome of combined light general anesthesia + high spinal block, with or without intrathecal morphine in patients undergoing cardiac-surgical procedures in our set up.

Null Hypothesis Addition of intrathecal morphine in high spinal anesthesia does not affect postoperative hemodynamics.

Aims and objectives A. Primary end point

1. To look for incidence of Vasoplegia (defined by MAP < 60mmHg with cardiac index > 2.2L/min/m2 or requirement of vasopressors to maintain the MAP > 60 mmHg in presence of cardiac index > 2.2L/min/m2) in the study groups.

B. Secondary end point 1. Mechanical ventilation duration, time to extubation, requirement of postoperative analgesia based on VAS, spirometry performance and incidence of awareness under anesthesia.

Materials and Methods After obtaining ethics committee approval and informed written consent of the patients, this study will be conducted in 60 adult patients with valvular heart disease and coronary artery disease of New York Heart Association class II-III aged 18 to 60 years undergoing elective cardiac surgery. All patients will receive their usual cardiovascular medications except angiotensin - converting enzyme inhibitors, digoxin and diuretics on the morning of surgery as per our institutional practice. On arrival inside operating room and after securing peripheral venous access with 16 G catheter, continuous monitoring will be instituted that will include 5-lead electrocardiogram, pulse oximetry, end-tidal capnometry, and invasive arterial blood pressure through a 20-G catheter inserted in a radial artery. A central venous catheter will be inserted before induction of anaesthesia under local anaesthesia and mild sedation with midazolam 0.04mg/kg body weight.

ANESTHESIA PROTOCOL:

Spinal anesthesia - All study patients will receive spinal anaesthesia prior to induction of GA. Patient will be placed in lateral position, parts painted and draped under strict aseptic precautions. Heavy bupivacaine 40 mg will be administered in all patients at the level of L2-3 or L3-4 intervertebral space in the Spinal group. Heavy bupivacaine (Anawin heavy 0.5%, Neon laboratories LTD, Thane, India) 40 mg mixed with preservative free morphine sulphate 250 mcg (VERMOR 15,Verve health care limited, Delhi, India) will be given in L2-3 or L3-4 space to all patients in the Opioid group. The patient will be then turned to supine position and a 30 degree Trendelenburg position will be maintained till sensory loss to a level of T1 is achieved. The sensory level will be assessed by loss of sensation to cold stimulation (Spirit swab), all the while administering 100% oxygen through a breathing system. Patient will receive 100% oxygen by mask for 10 minutes and in case of respiratory depression will be gently assisted in respiration. Once desired level is achieved, GA in both groups will be induced with midazolam 1-2 mg, ketamine 20-30 mg plus lignocaine 2mg/kg and propofol 20-40 mg titrated to maintain hemodynamics and to loss of eyelash reflex. Inj. Vecuronium bromide 0.1mg/kg will be used as muscle relaxant to facilitate tracheal intubation and lignocaine spray (LOX 10% spray, Neon laboratories LTD, Thane, India) will be used over vocal cords prior to intubation to blunt the sympathetic stimulation.

Subsequent anaesthesia will be maintained in all the patients in both the groups with isoflurane inhalation to maintain BIS values between 40-60 or end-tidal isoflurane of 1-MAC. Patients will be mechanically ventilated with 50% oxygen-air mixture and minute ventilation will be adjusted to achieve normocapnia till sternotomy. Vasoactive drug phenylephrine 100ug/ml will be prepared and boluses (1-2 ug/kg) given to all patients to maintain MAP > 60 mmHg (stable haemodynamics) on CPB. Normothermic CPB will be carried in all cases. Hematocrit of > 24% will be maintained in all patients on CPB. Total dose of phenylephrine received before and on bypass will be recorded in both the groups. Anesthesia and hemodynamics on cardiopulmonary bypass (CPB) will be maintained with isoflurane in oxygen-air mixture connected to the CPB machine and anesthesia post CPB period will be maintained with isoflurane in oxygen-air mixture. All patients will receive fentanyl 1ug/kg atleast 5-minutes before sternal closure.

Baseline pre-CPB TEE evaluation of LVOT diameter and LVOT area in ME-AV long axis view (average of three readings) will be recorded and used as a standard for subsequent calculation of cardiac output and cardiac index post-CPB and in ICU. Intra-operative TEE will be used to calculate the LVOT VTI (mean of three values) either in the transgastric long axis view or the deep transgastric long axis view (which ever gives better alignment) 15 minutes after separation from CPB and before transfer to ICU with simultaneous recording of systemic pressures (SBP,DBP and MAP). Vasoplegia in our study will be defined by mean arterial blood pressure < 60 mmHg with cardiac index ≥ 2.2 l/min/m2 or requirement for vasopressors to maintain MAP > 60 mmHg in presence of cardiac index ≥ 2.2 l/min/m2 65.

The mean of three reading taken five minutes apart before anaesthesia induction (prior to administration of spinal anaesthesia in spinal group) in both groups will be taken as baseline values.

Ionotropes will be used according to the underlying cardiac pathology. A combination of milrinone and norepinephrine will be used in patients with right ventricular dysfunction and pulmonary arterial hypertension ; a combination of dobutamine and norepinephrine/epinephrine will be used in patients with LV dysfunction ; in patients with biventricular dysfunction milrinone and norepinephrine/epinephrine will be used and low dose norepinephrine will be used in patients with diastolic dysfunction. Total dose of vasoactive drugs used in the postoperative period in the both the groups will be recorded in first 48 hours and analysed. In the ICU, following parameters will be recorded:

* Hemodynamic parameters (HR, SBP, DBP, MAP, CVP) will be recorded 4 hourly for 48 hours.
* Additional hemodynamic readings will be recorded at any point hemodynamic instability (defined by MAP < 60 mmHg).
* LVOT VTI will be measured in apical 5-chamber view and used to calculate SV. LVOT VTI derived will be multiplied with LVOT area (derived already on TEE) to calculate SV which will be multiplied by the HR of the patient at that point of time to calculate CO and CI every 4 hourly for 48 hours.
* Uniform rescue analgesia will be given to all the patients as per ICU protocol when the value on the Visual analog scale (VAS) is more than.

  . Postoperative Hb (gm/dl)
* Presence of residual sensory and motor blockade and occurrence of new onset motor blockade
* Duration of ventilation and time to extubation
* Record of complications (nausea,vomiting,pruritis) if any.
* Intra-operative awareness.
* Post-operative spirometry.

Statistical analysis

This will be taken as an open end, pilot feasibility study, that is, more of subjects will be added if the desired number (30) in each group is reached within less than the stipulated time period for thesis desertion submission.

Statistical analysis will be done using the SPSS software. All the parametric data such as hemodynamic parameters, time to extubation, and time to transfer to step down post anaesthesia care unit will be analysed using Unpaired t-tests. Chi-square (χ2) test will be used to analyse the requirement of vasoactive agents and the requirement of rescue analgesia. Residual sensory and motor blockade will be analysed using Mann-Whitney test

Proforma

Baseline demographics :Age(in years)/Sex (M/F)/Height (in meters)/Weight(in Kg's)/BSA(m2)/BMI (kg/m2).

Diagnosis :

Preoperative transthoracic echo findings:

LV EDD- LV ESD- LVEF-

Other findings:

Systemic illness:

Medication:

Laboratory results:

Hb: TLC: DLC: Platelet count:

PT: PTI: aPTT: INR:

Blood urea: Serum creatinine:

Serum bilirubin: SGOT/SGPT:

Time of spinal drug administration:

Time of tracheal intubation:

Time of incision:

Time of sternotomy:

LVOT Diameter = LVOT Area = Post-CPB LVEF TEMPERATURE MAINTAINED ON CPB = BASE EXCESS ON CPB = CPB TIME = AXC TIME = PONV = Y/N Hemodynamic Parameters: including HR,BP,CVP,LVOT VTI,CO,CI,LVEF and vasopressor dose will be recorded 4 hourly unto 48 hours in postoperative period.

Intravenous drugs given:All anesthetic drugs and ionotropes required to maintain stable hemodynamics during surgical procedure shall be recorded.

Requirement of vasoactive agent: over 48 hours in postoperative period shall be recorded

Time of shifting to PACU:

Postoperative parameters:

Requirement of analgesia- total dose of opioid and or non-opioid analgesics used over postoperative 48 hours shall be recorded Residual sensory blockade(Modified Bromage score): shall be recorded 4 hourly for 48 hours in postoperative period Residual motor blockade (Modified Bromage score):shall be recorded 4 hourly for 48 hours in postoperative period New onset motor blockade- Duration of ventilation- Time of extubation- Time of transfer to step down ICU- No of ICU hours- Post- extubation Volume achieved on incentive spirometry

1 hour 24 hours Awareness under Anaesthesia using Structured Brice and Bauer questionnaire shall also be recorded.

ELIGIBILITY:
Inclusion Criteria: - Adult patients with valvular heart disease and coronary artery disease of New York Heart Association class II-III aged 18 to 60 years undergoing elective cardiac surgery (Valve replacement/CABG).

Exclusion Criteria:

* • All the standard contraindications for spinal anaesthesia which includes local site infection, spinal deformity, coagulopathy (platelet count<80,000, INR>1.5) patients on anticoagulant medication continued upto the day of the surgery as per the third edition of the American Society of Regional Anesthesia and Pain Medicine Evidence-Based Guidelines (Regional Anesthesia in the Patient Receiving Antithrombotic or Thrombolytic Therapy)

  * Redo surgery/emergency surgeries.
  * Patients having co-morbidities such as obesity (BMI more than 30), COPD, asthma, that are likely to require prolonged post operative mechanical ventilation.
  * Total surgery time > 6 hours.
  * History of opioid drug abuse or patients on opioids for treatment of chronic pain.
  * Known or anticipated difficult airway

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
incidence of Vasoplegia | within 48 hours in post-operative period
  Vasoplegia (defined by MAP < 60mmHg with cardiac index > 2.2L/min/m2 or requirement of vasopressors to maintain the MAP > 60 mmHg in presence of cardiac index > 2.2L/min/m2)

SECONDARY OUTCOMES:
Mechanical ventilation duration. | post-operative 48 hours
  Hours of mechanical ventilation shall be noted for each patient and compared between the groups.
Time to extubation | within 48 hours in post-operative period
  Fast tracking (extubation within 6-8 hours of mechanical ventilation duration) or failure of fast tracking would be noted.
Requirement of postoperative analgesia based on VAS | upto 48 hours of postoperative period
  Rescue analgesic/s in the form of opioids/non-opioids will be administered if the VAS score exceeds 4 and note of drug and dose made.
Spirometry performance | Upto 48 postoperative hours.
  Two spirometry readings, one after extubation and another at 48 hours of postoperative period will be recorded
incidence of awareness under anesthesia | within 48 postoperative hours.
  Structured Brice and Bauer questionnaire shall be used to assess for intraoperative awareness.

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data will be furnished once asked for.

REFERENCES:
- [Derived] Bhat I, Arya VK, Mandal B, Jayant A, Dutta V, Rana SS. Postoperative hemodynamics after high spinal block with or without intrathecal morphine in cardiac surgical patients: a randomized-controlled trial. Can J Anaesth. 2021 Jun;68(6):825-834. doi: 10.1007/s12630-021-01937-z. Epub 2021 Feb 9. PMID 33564993